CLINICAL TRIAL: NCT05741580
Title: Evolution of Symptoms After Peri-urethral Bulk Agent Injection of Bulkamid® for Urinary Incontinence
Brief Title: Peri-urethral Bulk Agent Injection of Bulkamid®
Acronym: BULKIU
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5093; 69HCL22_1157 (Other: HCL)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence
Keywords: Bulkamid®; bulk agent; peri-urethral injection; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- peri-urethral bulk agent injection of Bulkamid® for urinary incontinence: patients who received a first injection of Bulkamid® in the context of urinary incontinence
  Interventions: Procedure: Evolution of symptoms

INTERVENTIONS:
Procedure: Evolution of symptoms — percentage of patients with improvement in their symptoms

SUMMARY:
There are currently different treatment options in the management of stress urinary incontinence according to the latest recommendations. Suburethral slings are currently considered the first surgical option due to an excellent cure rate of around 90%. Nevertheless, due to a risk of prosthetic complications and numerous current controversies over the placement of synthetic tissue, other therapeutic alternatives must be offered to patients.

Peri-urethral bulk agent injections have been used since 2006 in urinary incontinence and should be integrated into the therapeutic arsenal. This is a minimally invasive technique performed under local anesthesia on an outpatient basis. The mechanism of action is explained by better coaptation of the urethra and increased resistance to urine flow during the bladder filling phase. It also increases the strength of the striated sphincter thanks to a better arrangement of muscle fibers.

According to the European Association of Urology (EAU), the use of bulk agents is recommended for the management of urinary incontinence in elderly and/or frail patients whose comorbidities contraindicate surgical management. These peri-urethral injections can also be offered to patients with incontinence due to sphincter deficiency but also to young women with stress urinary incontinence who are ready to accept a partial improvement in their incontinence. The personal choice of the patient is currently a decisive factor for the implementation of a treatment for functional disorders and in particular for urinary incontinence.

ELIGIBILITY:
* Inclusion Criteria :

  * women over 18
  * patients who received a first peri-urethral injection of Bulkamid® in the context of urinary incontinence
  * intervention between September 2020 and November 2022
  * person having expressed his non-opposition
* Exclusion Criteria :

  * inability to understand the information given
  * person deprived of liberty
  * person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study concerns all patients who received a first peri-uthral injection of Bulkamid® in the context of urinary incontinence between September 2020 and November 2022.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evolution of symptoms | at 7 days after surgery
  percentage of patients with improvement in their symptoms on the PGI-I scale (score 1, 2, or 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie, HFME, Hospices Civils de Lyon, Bron, France